CLINICAL TRIAL: NCT01293188
Title: Observatory of Anticoagulation After Bioprosthetic Aortic Valve Replacement
Acronym: ARVA
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Bernard IUNG, Professor, French Cardiology Society
Other Study IDs: 10185
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Aortic Valve Disease
Keywords: Aortic Valve Replacement; Bioprosthetic
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biopresthetic aortic valve replacement.

SUMMARY:
The bioprosthetic aortic valve replacement is a frequent intervention because of the predominance of calcified aortic stenosis, which is the most common valvular disease, and aging of the population.

International guidelines recommend anticoagulant therapy during the 3 postoperative months, but the risk-benefit ratio of anticoagulation post-operatively is questioned because of the low level of evidence available studies and their sometimes conflicting conclusions.

Questionnaires sent to practitioners have highlighted discrepancies between common practices and recommendations.

However, there is no analysis of actual patterns of postoperative anticoagulation after aortic valve replacement with bioprosthesis.

The aim of the ARVA observatory is to establish a cohort of 600 patients enrolled in 3 months and had a bioprosthetic aortic valve replacement in one of the 22 surgical centers French.

DETAILED DESCRIPTION:
The study will include consecutive patients who agreed to participate in the study, which meet the criteria for inclusion, that is to say consecutive patients operated on by a bioprosthetic aortic valve replacement during the 3 months of inclusion. Patients will be included immediately after completion of aortic valve replacement.

The data will be entered directly by the referent of each center, based on data from the French Society of Cardiology accessible by Internet on a secure site.

The follow-up time will be 6 months

The incidence of thromboembolic complications and bleeding and mortality within 6 months will be analyzed in a standardized manner according to the recommendations on the analysis of morbidity and mortality after valve surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients operated on for single bioprosthetic aortic valve replacement during the study period:

  * with or without reinforcement
  * with or without associated CABG
  * with or without action on the ascending aorta
  * whether a first intervention or reoperation
* Patients who agreed to participate in the study

Exclusion Criteria:

* Replacement aortic valve homograft or autograft
* Surgical procedures on another valve (conservative or prosthetic replacement)
* Permanent Atrial Fibrillation
* Processing anticoagulant vitamin K-long course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with calcified aortic stenosis operated on for bioprosthetic aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 434 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mortality | 6 months

SECONDARY OUTCOMES:
Hemorragic and thrombo-embolitic complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Iung, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat Hospital, Paris, France

REFERENCES:
- [Background] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Background] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Background] Bonow RO, Carabello BA, Chatterjee K, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS; 2006 Writing Committee Members; American College of Cardiology/American Heart Association Task Force. 2008 Focused update incorporated into the ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 1998 Guidelines for the Management of Patients With Valvular Heart Disease): endorsed by the Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. Circulation. 2008 Oct 7;118(15):e523-661. doi: 10.1161/CIRCULATIONAHA.108.190748. Epub 2008 Sep 26. No abstract available. PMID 18820172
- [Background] Vahanian A, Baumgartner H, Bax J, Butchart E, Dion R, Filippatos G, Flachskampf F, Hall R, Iung B, Kasprzak J, Nataf P, Tornos P, Torracca L, Wenink A; Task Force on the Management of Valvular Hearth Disease of the European Society of Cardiology; ESC Committee for Practice Guidelines. Guidelines on the management of valvular heart disease: The Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology. Eur Heart J. 2007 Jan;28(2):230-68. doi: 10.1093/eurheartj/ehl428. Epub 2007 Jan 26. No abstract available. PMID 17259184
- [Background] Salem DN, O'Gara PT, Madias C, Pauker SG. Valvular and structural heart disease: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):593S-629S. doi: 10.1378/chest.08-0724. PMID 18574274
- [Background] Dunning J, Versteegh M, Fabbri A, Pavie A, Kolh P, Lockowandt U, Nashef SA; EACTS Audit and Guidelines Committee. Guideline on antiplatelet and anticoagulation management in cardiac surgery. Eur J Cardiothorac Surg. 2008 Jul;34(1):73-92. doi: 10.1016/j.ejcts.2008.02.024. Epub 2008 Mar 28. PMID 18375137
- [Background] Colli A, Verhoye JP, Heijmen R, Strauch JT, Hyde JA, Pagano D, Antunes M, Koertke H, Ohri SK, Bail DH, Leprince P, Van Straten BH, Gherli T; ACTION Registry Investigators. Antithrombotic therapy after bioprosthetic aortic valve replacement: ACTION Registry survey results. Eur J Cardiothorac Surg. 2008 Apr;33(4):531-6. doi: 10.1016/j.ejcts.2007.12.019. Epub 2008 Jan 18. PMID 18203613
- [Background] Vaughan P, Waterworth PD. An audit of anticoagulation practice among UK cardiothoracic consultant surgeons following valve replacement/repair. J Heart Valve Dis. 2005 Sep;14(5):576-82. PMID 16245494
- [Background] Aramendi JI, Mestres CA, Martinez-Leon J, Campos V, Munoz G, Navas C. Triflusal versus oral anticoagulation for primary prevention of thromboembolism after bioprosthetic valve replacement (trac): prospective, randomized, co-operative trial. Eur J Cardiothorac Surg. 2005 May;27(5):854-60. doi: 10.1016/j.ejcts.2004.12.064. PMID 15848326
- [Background] Gherli T, Colli A, Fragnito C, Nicolini F, Borrello B, Saccani S, D'Amico R, Beghi C. Comparing warfarin with aspirin after biological aortic valve replacement: a prospective study. Circulation. 2004 Aug 3;110(5):496-500. doi: 10.1161/01.cir.0000137122.95108.52. PMID 15289387
- [Background] Heras M, Chesebro JH, Fuster V, Penny WJ, Grill DE, Bailey KR, Danielson GK, Orszulak TA, Pluth JR, Puga FJ, et al. High risk of thromboemboli early after bioprosthetic cardiac valve replacement. J Am Coll Cardiol. 1995 Apr;25(5):1111-9. doi: 10.1016/0735-1097(94)00563-6. PMID 7897124
- [Background] Orszulak TA, Schaff HV, Mullany CJ, Anderson BJ, Ilstrup DM, Puga FJ, Danielson GK. Risk of thromboembolism with the aortic Carpentier-Edwards bioprosthesis. Ann Thorac Surg. 1995 Feb;59(2):462-8. doi: 10.1016/0003-4975(94)00862-2. PMID 7847967
- [Background] Moinuddeen K, Quin J, Shaw R, Dewar M, Tellides G, Kopf G, Elefteriades J. Anticoagulation is unnecessary after biological aortic valve replacement. Circulation. 1998 Nov 10;98(19 Suppl):II95-8; discussion II98-9. PMID 9852888
- [Background] Blair KL, Hatton AC, White WD, Smith LR, Lowe JE, Wolfe WG, Young WG, Oldham HN, Douglas JM Jr, Glower DD. Comparison of anticoagulation regimens after Carpentier-Edwards aortic or mitral valve replacement. Circulation. 1994 Nov;90(5 Pt 2):II214-9. PMID 7955256
- [Background] Sundt TM, Zehr KJ, Dearani JA, Daly RC, Mullany CJ, McGregor CG, Puga FJ, Orszulak TA, Schaff HV. Is early anticoagulation with warfarin necessary after bioprosthetic aortic valve replacement? J Thorac Cardiovasc Surg. 2005 May;129(5):1024-31. doi: 10.1016/j.jtcvs.2004.11.028. PMID 15867776
- [Background] Brueck M, Kramer W, Vogt P, Steinert N, Roth P, Gorlach G, Schonburg M, Heidt MC. Antiplatelet therapy early after bioprosthetic aortic valve replacement is unnecessary in patients without thromboembolic risk factors. Eur J Cardiothorac Surg. 2007 Jul;32(1):108-12. doi: 10.1016/j.ejcts.2007.03.031. Epub 2007 Apr 20. PMID 17449264
- [Background] Iung B. Management of the elderly patient with aortic stenosis. Heart. 2008 Apr;94(4):519-24. doi: 10.1136/hrt.2007.122804. No abstract available. PMID 18347382
- [Background] Akins CW, Miller DC, Turina MI, Kouchoukos NT, Blackstone EH, Grunkemeier GL, Takkenberg JJ, David TE, Butchart EG, Adams DH, Shahian DM, Hagl S, Mayer JE, Lytle BW; Councils of the American Association for Thoracic Surgery; Society of Thoracic Surgeons; European Assoication for Cardio-Thoracic Surgery; Ad Hoc Liaison Committee for Standardizing Definitions of Prosthetic Heart Valve Morbidity. Guidelines for reporting mortality and morbidity after cardiac valve interventions. J Thorac Cardiovasc Surg. 2008 Apr;135(4):732-8. doi: 10.1016/j.jtcvs.2007.12.002. No abstract available. PMID 18374749